CLINICAL TRIAL: NCT03353311
Title: ERAS Lazio Network Clinical Registry
Acronym: ENeRgy
Status: Completed | Type: Observational
Sponsor: PERSIANI ROBERTO (Other)
Collaborators: Azienda Ospedaliera "Sant'Andrea" (Other); Policlinico Casilino ASL RMB (Other); San Giovanni Addolorata Hospital (Other); Campus Bio-Medico University (Other); Ospedale San Paolo Civitavecchia (Unknown); Ospedale Cristo Re - Roma (Unknown); S.Eugenio Hospital (Other)
Responsible Party: Sponsor-Investigator, PERSIANI ROBERTO, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Organization: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Other Study IDs: FPAG001
Record Dates: First submitted 2017-11-14; First posted 2017-11-27 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Colon Cancer; Diverticulum, Colon
Keywords: ERAS; Fast-track; colorectal surgery; immuno-nutrition
MeSH Terms: conditions — Colonic Neoplasms; Diverticulum, Colon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Enhanced Recovery After Surgery: Patients undergoing elective colorectal surgical resection for benign/malignant disease.
  A multidisciplinary validated approach based on 24 items including Preadmission information, education and counselling Preoperative optimization (increasing exercise, stop smoking and alcohol consumption should 4 weeks before surgery) No preoperative bowel preparation Use of preoperative carbohydrate drinks Pre-anesthetic medication Prophylaxis against thromboembolism Antimicrobial prophylaxis and skin preparation Standard anesthetic protocol for rapid awakening PONV Mini-invasive surgery No nasogastric dreinage Prevention of intraoperative hypothermia Perioperative fluid management No drains in the peritoneal cavity after colonic anastomosis Early remouval of urinary drainage (24-48 hrs) Prevention of postoperative ileus (including use of postoperative laxatives) Postoperative analgesia Perioperative nutritional care Postoperative control of glucose Early mobilization Auditing

SUMMARY:
Enhanced recovery after surgery (ERAS) protocols are programs aiming to implement patients recovery following surgical procedures developed about 25 years ago. ERAS protocols are based on a multi-disciplinary approach encompassing surgery, anesthesiology, nutrition and nursing; each specialty has to fulfill a number of items which have been demonstrated to reduce morbidity rates, hospital stay and to implement functional recovery comparing standard approach. Accordingly, ERAS society developed a Guidelines for a number of procedures, including colorectal.

The aim of this study is to evaluate the adherence over the last years to these protocols in eight Department of Surgery in Rome in a series of colorectal cancer patients.

Secondary aims are to investigate the correlation of the items adherence with surgical outcome and to establish a network of hospitals aiming to promote ERAS approach on a regional base.

DETAILED DESCRIPTION:
Background. The acronym ERAS (Enhanced Recovery After Surgery) refers to a patient-centered, evidence-based multi-disciplinary protocol designed to implement perioperative operation, reduce surgical trauma, and facilitate recovery of physiological functions aiming to an early hospital discharge.

Usually ERAS protocols give a continuum of care starting at home (pre-hospital/pre-admission phase) to continue in followed by the pre-/ intra-/ and post-operative phases.

ERAS includes a wide range of disciplines and specialists, which focus on the needs of the patient in order to improve support by facilitating his return home.

The first author to introduce the fast-track term in rectal surgery was Prof. Henrik Kehlet in the mid-1990s, proposing a multi-modal rehabilitation program aimed to reduce post-surgical stress response, morbidity, mortality and postoperative hospitalization. Since then, a number of studies were conducted leading to the first ERAS protocol; since then, these protocols were reviewed on a regular basis, the last time in 2017 and included in the guidelines by the ERAS society (http://www.erassociety.org).

Currently, it is widely demonstrated that, comparing to a traditional approach, ERAS is associated with a significant reduction in morbidity, days of hospitalization, mortality, implementing early postoperative recovery with a consequent reduction of the costs, without compromising patient safety.

In particular, ERAS for colorectal surgery, includes 24 demonstrated multi-disciplinary.

Aims. the investigators aim to evaluate the adherence to the individual items and the short-term outcomes (postoperative hospitalization, complication rates within 30 days of intervention, re-intervention) in a consecutive series of patients undergoing colorectal resection, in eight centers in the Lazio region, treated according to the ERAS protocol.

Secondary aims are to investigate the correlation of the items adherence with surgical outcome and to establish a network of hospitals aiming to promote ERAS approach on a regional base.

Design. This is a no-profit, spontaneous, observational, non-intervention Audit collecting data in eight surgical Departments based in Lazio region, since September 2014 to October 2017. Each participating center will be depositary of its own data.

Participating Centers.

1. UOC General Surgery 1, Fondazione Policlinico Universitario "A. Gemelli ", Rome (Coordinator) -
2. Department of Surgery, S. Eugenio Hospital, Rome
3. UOD Week-Day Surgery, St. Andrea Hospital, Rome
4. UOC General Surgery, Polyclinic University Bio-Medical Campus, Rome
5. UO General and Urgent Surgery, Policlinico Casilino Hospital, Rome
6. UOC Surgery, San Paolo Hospital, Civitavechia (RM)
7. UOC General Surgery, Cristo Re Hospital, Rome
8. UOSD Robotic Surgery for General Surgery, San Giovanni-Addolorata Hospital, Rome

Data Collection. Each center will collect the data in a homogeneous Database. The data will be collected in anonymous form and will be aimed at the definition of:

1. Duration of postoperative stay
2. Short-term morbidity rate (within 30 days) according to Clavien-Dindo classification
3. Re-intervention rate (within 30 days)
4. Hospital readmission (within 30 days)

f. Adherence rate to items of the series All data will be treated sensibly; each patient will be recorded with a sequential center-specific code. For all new patients and for patients seen in follow-up visits, the specific informed consent of the study will be compiled.

Statistical analysis. Categorical variables will be presented as rate and percentages, the continuous variables as mean, median, and standard deviation.

A logistic regression will also be performed, computing items as co-variates, with the end-point of post-operative morbidity and hospital stay.

Sample Size Calculation: 1000 patients, calculated on the basis of the annual case of each participating center.

For the conduct and management of this observational study no additional cost will be charged on NHS funds.

ELIGIBILITY:
Inclusion Criteria:

* Elective colorectal surgical resection
* Open and Laparoscopic Suregry
* Benign/malignant disease
* independently from age, sex,

Exclusion Criteria:

Emergency colorectal resections

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Open or laparoscopic colorectal surgical resection for a benign/malignant disease independently from patients age or sex
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Adherance to ERAS protocol | 36 months
  Number of items included in the ERAS protocols that were applied in each centre

SECONDARY OUTCOMES:
Number of items of the ERAS protol correlated wih adverse events as described by the Clavien Dindo Classification and with a longer hospital stay | 36 months
  Multivariate analysis to relate ERAS items to morbidity or a longer hospital stay (>mean values)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Unversitario Agostino Gemelli, Roma, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared

REFERENCES:
- [Background] Bardram L, Funch-Jensen P, Jensen P, Crawford ME, Kehlet H. Recovery after laparoscopic colonic surgery with epidural analgesia, and early oral nutrition and mobilisation. Lancet. 1995 Mar 25;345(8952):763-4. doi: 10.1016/s0140-6736(95)90643-6. PMID 7891489
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] Fearon KC, Ljungqvist O, Von Meyenfeldt M, Revhaug A, Dejong CH, Lassen K, Nygren J, Hausel J, Soop M, Andersen J, Kehlet H. Enhanced recovery after surgery: a consensus review of clinical care for patients undergoing colonic resection. Clin Nutr. 2005 Jun;24(3):466-77. doi: 10.1016/j.clnu.2005.02.002. Epub 2005 Apr 21. PMID 15896435
- [Background] Lassen K, Soop M, Nygren J, Cox PB, Hendry PO, Spies C, von Meyenfeldt MF, Fearon KC, Revhaug A, Norderval S, Ljungqvist O, Lobo DN, Dejong CH; Enhanced Recovery After Surgery (ERAS) Group. Consensus review of optimal perioperative care in colorectal surgery: Enhanced Recovery After Surgery (ERAS) Group recommendations. Arch Surg. 2009 Oct;144(10):961-9. doi: 10.1001/archsurg.2009.170. PMID 19841366
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, Macfie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):259-84. doi: 10.1007/s00268-012-1772-0. No abstract available. PMID 23052794
- [Background] Kehlet H, Wilmore DW. Evidence-based surgical care and the evolution of fast-track surgery. Ann Surg. 2008 Aug;248(2):189-98. doi: 10.1097/SLA.0b013e31817f2c1a. PMID 18650627
- [Background] Wind J, Polle SW, Fung Kon Jin PH, Dejong CH, von Meyenfeldt MF, Ubbink DT, Gouma DJ, Bemelman WA; Laparoscopy and/or Fast Track Multimodal Management Versus Standard Care (LAFA) Study Group; Enhanced Recovery after Surgery (ERAS) Group. Systematic review of enhanced recovery programmes in colonic surgery. Br J Surg. 2006 Jul;93(7):800-9. doi: 10.1002/bjs.5384. PMID 16775831
- [Background] Eskicioglu C, Forbes SS, Aarts MA, Okrainec A, McLeod RS. Enhanced recovery after surgery (ERAS) programs for patients having colorectal surgery: a meta-analysis of randomized trials. J Gastrointest Surg. 2009 Dec;13(12):2321-9. doi: 10.1007/s11605-009-0927-2. Epub 2009 May 21. PMID 19459015
- [Background] Kondrup J, Allison SP, Elia M, Vellas B, Plauth M; Educational and Clinical Practice Committee, European Society of Parenteral and Enteral Nutrition (ESPEN). ESPEN guidelines for nutrition screening 2002. Clin Nutr. 2003 Aug;22(4):415-21. doi: 10.1016/s0261-5614(03)00098-0. PMID 12880610
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673
- [Background] Awad S, Lobo DN. What's new in perioperative nutritional support? Curr Opin Anaesthesiol. 2011 Jun;24(3):339-48. doi: 10.1097/ACO.0b013e328345865e. PMID 21451404
- [Background] Ali Abdelhamid Y, Chapman MJ, Deane AM. Peri-operative nutrition. Anaesthesia. 2016 Jan;71 Suppl 1:9-18. doi: 10.1111/anae.13310. PMID 26620142
- [Background] Black PR, Brooks DC, Bessey PQ, Wolfe RR, Wilmore DW. Mechanisms of insulin resistance following injury. Ann Surg. 1982 Oct;196(4):420-35. doi: 10.1097/00000658-198210000-00005. PMID 6751244
- [Background] Nygren J, Thorell A, Ljungqvist O. Preoperative oral carbohydrate nutrition: an update. Curr Opin Clin Nutr Metab Care. 2001 Jul;4(4):255-9. doi: 10.1097/00075197-200107000-00002. PMID 11458017
- [Background] Jung B, Pahlman L, Nystrom PO, Nilsson E; Mechanical Bowel Preparation Study Group. Multicentre randomized clinical trial of mechanical bowel preparation in elective colonic resection. Br J Surg. 2007 Jun;94(6):689-95. doi: 10.1002/bjs.5816. PMID 17514668
- [Background] Contant CM, Hop WC, van't Sant HP, Oostvogel HJ, Smeets HJ, Stassen LP, Neijenhuis PA, Idenburg FJ, Dijkhuis CM, Heres P, van Tets WF, Gerritsen JJ, Weidema WF. Mechanical bowel preparation for elective colorectal surgery: a multicentre randomised trial. Lancet. 2007 Dec 22;370(9605):2112-7. doi: 10.1016/S0140-6736(07)61905-9. PMID 18156032
- [Background] Noblett SE, Watson DS, Huong H, Davison B, Hainsworth PJ, Horgan AF. Pre-operative oral carbohydrate loading in colorectal surgery: a randomized controlled trial. Colorectal Dis. 2006 Sep;8(7):563-9. doi: 10.1111/j.1463-1318.2006.00965.x. PMID 16919107
- [Background] Slim K, Vicaut E, Panis Y, Chipponi J. Meta-analysis of randomized clinical trials of colorectal surgery with or without mechanical bowel preparation. Br J Surg. 2004 Sep;91(9):1125-30. doi: 10.1002/bjs.4651. PMID 15449262
- [Background] Wille-Jorgensen P, Guenaga KF, Castro AA, Matos D. Clinical value of preoperative mechanical bowel cleansing in elective colorectal surgery: a systematic review. Dis Colon Rectum. 2003 Aug;46(8):1013-20. doi: 10.1007/s10350-004-7274-x. PMID 12907890
- [Background] Platell C, Hall J. What is the role of mechanical bowel preparation in patients undergoing colorectal surgery? Dis Colon Rectum. 1998 Jul;41(7):875-82; discussion 882-3. doi: 10.1007/BF02235369. PMID 9678373
- [Background] Guenaga KF, Matos D, Castro AA, Atallah AN, Wille-Jorgensen P. Mechanical bowel preparation for elective colorectal surgery. Cochrane Database Syst Rev. 2003;(2):CD001544. doi: 10.1002/14651858.CD001544. PMID 12804412
- [Background] Kwon S, Meissner M, Symons R, Steele S, Thirlby R, Billingham R, Flum DR; Surgical Care and Outcomes Assessment Program Collaborative. Perioperative pharmacologic prophylaxis for venous thromboembolism in colorectal surgery. J Am Coll Surg. 2011 Nov;213(5):596-603, 603.e1. doi: 10.1016/j.jamcollsurg.2011.07.015. Epub 2011 Aug 25. PMID 21871823
- [Background] van Dongen CJ, MacGillavry MR, Prins MH. Once versus twice daily LMWH for the initial treatment of venous thromboembolism. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD003074. doi: 10.1002/14651858.CD003074.pub2. PMID 16034885
- [Background] Rasmussen MS, Jorgensen LN, Wille-Jorgensen P. Prolonged thromboprophylaxis with low molecular weight heparin for abdominal or pelvic surgery. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD004318. doi: 10.1002/14651858.CD004318.pub2. PMID 19160234
- [Background] Song F, Glenny AM. Antimicrobial prophylaxis in colorectal surgery: a systematic review of randomized controlled trials. Br J Surg. 1998 Sep;85(9):1232-41. doi: 10.1046/j.1365-2168.1998.00883.x. PMID 9752867
- [Background] Bratzler DW, Houck PM; Surgical Infection Prevention Guidelines Writers Workgroup; American Academy of Orthopaedic Surgeons; American Association of Critical Care Nurses; American Association of Nurse Anesthetists; American College of Surgeons; American College of Osteopathic Surgeons; American Geriatrics Society; American Society of Anesthesiologists; American Society of Colon and Rectal Surgeons; American Society of Health-System Pharmacists; American Society of PeriAnesthesia Nurses; Ascension Health; Association of periOperative Registered Nurses; Association for Professionals in Infection Control and Epidemiology; Infectious Diseases Society of America; Medical Letter; Premier; Society for Healthcare Epidemiology of America; Society of Thoracic Surgeons; Surgical Infection Society. Antimicrobial prophylaxis for surgery: an advisory statement from the National Surgical Infection Prevention Project. Clin Infect Dis. 2004 Jun 15;38(12):1706-15. doi: 10.1086/421095. Epub 2004 May 26. PMID 15227616
- [Background] Steinberg JP, Braun BI, Hellinger WC, Kusek L, Bozikis MR, Bush AJ, Dellinger EP, Burke JP, Simmons B, Kritchevsky SB; Trial to Reduce Antimicrobial Prophylaxis Errors (TRAPE) Study Group. Timing of antimicrobial prophylaxis and the risk of surgical site infections: results from the Trial to Reduce Antimicrobial Prophylaxis Errors. Ann Surg. 2009 Jul;250(1):10-6. doi: 10.1097/SLA.0b013e3181ad5fca. PMID 19561486
- [Background] Fujita S, Saito N, Yamada T, Takii Y, Kondo K, Ohue M, Ikeda E, Moriya Y. Randomized, multicenter trial of antibiotic prophylaxis in elective colorectal surgery: single dose vs 3 doses of a second-generation cephalosporin without metronidazole and oral antibiotics. Arch Surg. 2007 Jul;142(7):657-61. doi: 10.1001/archsurg.142.7.657. PMID 17638804
- [Background] Walker KJ, Smith AF. Premedication for anxiety in adult day surgery. Cochrane Database Syst Rev. 2009 Oct 7;2009(4):CD002192. doi: 10.1002/14651858.CD002192.pub2. PMID 19821294
- [Background] Levy BF, Scott MJ, Fawcett WJ, Day A, Rockall TA. Optimizing patient outcomes in laparoscopic surgery. Colorectal Dis. 2011 Nov;13 Suppl 7:8-11. doi: 10.1111/j.1463-1318.2011.02770.x. PMID 22098510
- [Background] Punjasawadwong Y, Boonjeungmonkol N, Phongchiewboon A. Bispectral index for improving anaesthetic delivery and postoperative recovery. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD003843. doi: 10.1002/14651858.CD003843.pub2. PMID 17943802
- [Background] Varadhan KK, Lobo DN. A meta-analysis of randomised controlled trials of intravenous fluid therapy in major elective open abdominal surgery: getting the balance right. Proc Nutr Soc. 2010 Nov;69(4):488-98. doi: 10.1017/S0029665110001734. Epub 2010 Jun 2. PMID 20515521
- [Background] Bundgaard-Nielsen M, Secher NH, Kehlet H. 'Liberal' vs. 'restrictive' perioperative fluid therapy--a critical assessment of the evidence. Acta Anaesthesiol Scand. 2009 Aug;53(7):843-51. doi: 10.1111/j.1399-6576.2009.02029.x. Epub 2009 Jun 10. PMID 19519723
- [Background] Cheatham ML, Chapman WC, Key SP, Sawyers JL. A meta-analysis of selective versus routine nasogastric decompression after elective laparotomy. Ann Surg. 1995 May;221(5):469-76; discussion 476-8. doi: 10.1097/00000658-199505000-00004. PMID 7748028
- [Background] Nelson R, Tse B, Edwards S. Systematic review of prophylactic nasogastric decompression after abdominal operations. Br J Surg. 2005 Jun;92(6):673-80. doi: 10.1002/bjs.5090. PMID 15912492
- [Background] Rao W, Zhang X, Zhang J, Yan R, Hu Z, Wang Q. The role of nasogastric tube in decompression after elective colon and rectum surgery: a meta-analysis. Int J Colorectal Dis. 2011 Apr;26(4):423-9. doi: 10.1007/s00384-010-1093-4. Epub 2010 Nov 24. PMID 21107848
- [Background] Camus Y, Delva E, Cohen S, Lienhart A. The effects of warming intravenous fluids on intraoperative hypothermia and postoperative shivering during prolonged abdominal surgery. Acta Anaesthesiol Scand. 1996 Aug;40(7):779-82. doi: 10.1111/j.1399-6576.1996.tb04532.x. PMID 8874562
- [Background] Galvao CM, Marck PB, Sawada NO, Clark AM. A systematic review of the effectiveness of cutaneous warming systems to prevent hypothermia. J Clin Nurs. 2009 Mar;18(5):627-36. doi: 10.1111/j.1365-2702.2008.02668.x. PMID 19239533
- [Background] Karanicolas PJ, Smith SE, Kanbur B, Davies E, Guyatt GH. The impact of prophylactic dexamethasone on nausea and vomiting after laparoscopic cholecystectomy: a systematic review and meta-analysis. Ann Surg. 2008 Nov;248(5):751-62. doi: 10.1097/SLA.0b013e3181856024. PMID 18948802
- [Background] Habib AS, El-Moalem HE, Gan TJ. The efficacy of the 5-HT3 receptor antagonists combined with droperidol for PONV prophylaxis is similar to their combination with dexamethasone. A meta-analysis of randomized controlled trials. Can J Anaesth. 2004 Apr;51(4):311-9. doi: 10.1007/BF03018234. PMID 15064259
- [Background] Zafar N, Davies R, Greenslade GL, Dixon AR. The evolution of analgesia in an 'accelerated' recovery programme for resectional laparoscopic colorectal surgery with anastomosis. Colorectal Dis. 2010 Feb;12(2):119-24. doi: 10.1111/j.1463-1318.2009.01768.x. Epub 2009 Jan 16. PMID 19207712
- [Background] Gustafsson UO, Thorell A, Soop M, Ljungqvist O, Nygren J. Haemoglobin A1c as a predictor of postoperative hyperglycaemia and complications after major colorectal surgery. Br J Surg. 2009 Nov;96(11):1358-64. doi: 10.1002/bjs.6724. PMID 19847870
- [Background] Nygren J, Soop M, Thorell A, Hausel J, Ljungqvist O; ERAS Group. An enhanced-recovery protocol improves outcome after colorectal resection already during the first year: a single-center experience in 168 consecutive patients. Dis Colon Rectum. 2009 May;52(5):978-85. doi: 10.1007/DCR.0b013e31819f1416. PMID 19502866
- [Background] Hannemann P, Lassen K, Hausel J, Nimmo S, Ljungqvist O, Nygren J, Soop M, Fearon K, Andersen J, Revhaug A, von Meyenfeldt MF, Dejong CH, Spies C. Patterns in current anaesthesiological peri-operative practice for colonic resections: a survey in five northern-European countries. Acta Anaesthesiol Scand. 2006 Oct;50(9):1152-60. doi: 10.1111/j.1399-6576.2006.01121.x. Epub 2006 Aug 25. PMID 16939479
- [Background] Lewis SJ, Egger M, Sylvester PA, Thomas S. Early enteral feeding versus "nil by mouth" after gastrointestinal surgery: systematic review and meta-analysis of controlled trials. BMJ. 2001 Oct 6;323(7316):773-6. doi: 10.1136/bmj.323.7316.773. PMID 11588077
- [Background] Han-Geurts IJ, Hop WC, Kok NF, Lim A, Brouwer KJ, Jeekel J. Randomized clinical trial of the impact of early enteral feeding on postoperative ileus and recovery. Br J Surg. 2007 May;94(5):555-61. doi: 10.1002/bjs.5753. PMID 17443854
- [Background] Vlug MS, Wind J, Hollmann MW, Ubbink DT, Cense HA, Engel AF, Gerhards MF, van Wagensveld BA, van der Zaag ES, van Geloven AA, Sprangers MA, Cuesta MA, Bemelman WA; LAFA study group. Laparoscopy in combination with fast track multimodal management is the best perioperative strategy in patients undergoing colonic surgery: a randomized clinical trial (LAFA-study). Ann Surg. 2011 Dec;254(6):868-75. doi: 10.1097/SLA.0b013e31821fd1ce. PMID 21597360
- [Background] Houborg KB, Jensen MB, Hessov I, Laurberg S. Little effect of physical training on body composition and nutritional intake following colorectal surgery--a randomised placebo-controlled trial. Eur J Clin Nutr. 2005 Aug;59(8):969-77. doi: 10.1038/sj.ejcn.1602198. PMID 15970946